CLINICAL TRIAL: NCT01701895
Title: CID 1213 - Assessing Short and Long Term Compliance With Caloric Intake in HIV Positive Women After Switching to Fixed Dose Combination of Rilpivirine, Emtricitabine and Tenofovir DF
Brief Title: Assessing Short and Long Term Compliance With Caloric Intake in HIV Positive Women Taking Complera
Status: Completed | Type: Observational
Sponsor: Prema Menezes, PhD, PA-C (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Prema Menezes, PhD, PA-C, Clinical Assistant Professor of Medicine, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: CID 1213 - IRB 12-1550
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: HIV-1 Infection
Keywords: Complera; short-term; long-term; compliance; caloric; intake; HIV; positive; women
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to evaluate how easy it is for female HIV- positive subjects taking Complera to comply with the dietary requirement using a food diary in the short term (4 weeks) and long term (24 weeks and 48 weeks) and to determine association between calorie intake and virologic suppression. A secondary goal of the study is to evaluate subjects' attitudes towards contraception.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection documented by HIV serology or detectable viral load at any point prior to study entry or other documentation confirming HIV infection. If no documentation is available to confirm HIV infection, a rapid test may be performed to document HIV infection.
2. HIV+ female ≥18 years old and obtaining care at UNC Health Care Infectious Diseases Clinic, Wake County Human Services Clinic, or Durham County Early Intervention Clinic. Patients receiving care at other clinics may be entered with approval of the study team.
3. HIV viral load (VL) < 50 copies/ml as measured by any FDA-approved test for quantifying HIV-1 RNA during the six months prior to study entry (PSE). The timing of the viral load may be longer than 6 months depending on the schedule of the last clinic visit attended by the subject. The intent of the protocol was to assess viral load status at the previous clinic visit which may occur at an interval longer than six months due to the scheduling constraints of the UNC Infectious Diseases clinic. Viral loads drawn > than 6 months (but not > 8 months) prior to the study entry visit are acceptable. A single "blip" of > 50 and < 200 copies/ml is permissible provided the most recent VL is <50 copies/ml.
4. No documented resistance to FTC, TDF or rilpivirine. Note: genotyping will not be performed on study. Subjects with no historical genotype will be considered to have no documented resistance.
5. Able and willing to provide informed consent.
6. In the opinion of the investigator, able to comply with study medication and procedures, including ability to complete food diary.
7. Willing to receive monthly phone calls.
8. Agreement between ID clinic provider and study team that clinical monitoring and care of patient will reside with the ID clinic provider. The study responsibility is limited to providing 48 weeks of Complera.

Exclusion Criteria:

1. Any condition which, in the opinion of the investigator, would be likely to interfere with ability to take the study medications appropriately and comply with the study protocol.
2. Current active illness requiring systemic treatment and/or hospitalization until the individual completes therapy or, in the opinion of the investigator, is clinically stable on therapy for at least 7 days prior to study entry.
3. Acute viral hepatitis.
4. Known allergy/hypersensitivity to components of the study drugs or their formulations.
5. Current or expected use of medication on the prohibited medication list.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive females ≥ 18 years of age who are currently on Complera with suppressed viral load (VL) defined as having VL <50 copies/ml in the 6 months prior to study entry and no known resistance to FTC, TDF, or rilpivirine. Subjects may or may not be of child bearing potential.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Compliance with meal instruction | once per month over 48 weeks
  Compliance will be assessed monthly by a subject-completed food diary and phone assessments.

SECONDARY OUTCOMES:
Evaluation of subjects' attitudes toward contraception | up to 48 weeks
  Subjects are questioned about their contraceptive choices.
Association between caloric intake and virologic suppression | up to 48 weeks
Assessment of medication adherence | up to 48 weeks
  Subjects will self-report adherence on a visual analog scale.

OTHER OUTCOMES:
Measurement of change in fasting lipids | Week 48
Measurement of change in fasting lipids | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Prema Menezes, PhD, PA-C, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Panel on Antiretroviral Guidelines for Adults and Adolescents. Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. Department of Health and Human Services. January 10, 2011; 1-166. Available at http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL.pdf. Accessed 20Jun2011
- [Background] Bartlett JA, Fath MJ, Demasi R, Hermes A, Quinn J, Mondou E, Rousseau F. An updated systematic overview of triple combination therapy in antiretroviral-naive HIV-infected adults. AIDS. 2006 Oct 24;20(16):2051-64. doi: 10.1097/01.aids.0000247578.08449.ff. PMID 17053351
- [Background] El-Ibiary SY, Cocohoba JM. Effects of HIV antiretrovirals on the pharmacokinetics of hormonal contraceptives. Eur J Contracept Reprod Health Care. 2008 Jun;13(2):123-32. doi: 10.1080/13625180701829952. PMID 18465473
- [Background] Sekar V, Ryan R, Schaible D, et al Pharmacokinetic profile of darunavir co-administered with low-dose ritonavir in treatment-experienced women and men with HIV infection: 4-week analysis in a substudy of the GRACE (Gender, Race, And Clinical Experience) study. 9th International Workshop on Clinical Pharmacology of HIV Therapy. April 7-9, 2008. New Orleans. Abstract O16
- [Background] Umeh O, Currier J, Park JG et al. Sex differences in lopinavir/ritonavir soft gel capsule pharmacokinetics among HIV infected females and males. Conference on Retroviruses and Opportunistic Infections. February 3-6,2008, Boston, Massachusetts Abstract 786
- [Background] Ford N, Lee J, Andrieux-Meyer I, Calmy A. Safety, efficacy, and pharmacokinetics of rilpivirine: systematic review with an emphasis on resource-limited settings. HIV AIDS (Auckl). 2011;3:35-44. doi: 10.2147/HIV.S14559. Epub 2011 Apr 28. PMID 22096405
- [Background] Cohen C, Molina JM, Cahn P et al, Pooled 48 week efficacy and safety results from ECHO and THRIVE, two double blind randomized Phase III trials comparing TMC 278 vs. efavirenz in treatment naïve HIV-1 infected patients. HIV DART 2010 Abstract 45
- [Background] Hodder SL, Mounzer K, Dejesus E, Ebrahimi R, Grimm K, Esker S, Ecker J, Farajallah A, Flaherty JF; AI266073 Study Group. Patient-reported outcomes in virologically suppressed, HIV-1-Infected subjects after switching to a simplified, single-tablet regimen of efavirenz, emtricitabine, and tenofovir DF. AIDS Patient Care STDS. 2010 Feb;24(2):87-96. doi: 10.1089/apc.2009.0259. PMID 20156091
- [Background] Walsh JC, Mandalia S, Gazzard BG. Responses to a 1 month self-report on adherence to antiretroviral therapy are consistent with electronic data and virological treatment outcome. AIDS. 2002 Jan 25;16(2):269-77. doi: 10.1097/00002030-200201250-00017. PMID 11807312
- [Background] Giordano TP, Guzman D, Clark R, Charlebois ED, Bangsberg DR. Measuring adherence to antiretroviral therapy in a diverse population using a visual analogue scale. HIV Clin Trials. 2004 Mar-Apr;5(2):74-9. doi: 10.1310/JFXH-G3X2-EYM6-D6UG. PMID 15116282
- [Background] Prins M, Meyer L, Hessol NA. Sex and the course of HIV infection in the pre- and highly active antiretroviral therapy eras. AIDS. 2005 Mar 4;19(4):357-70. doi: 10.1097/01.aids.0000161765.75663.27. PMID 15750389
- [Background] Justice AC, Holmes W, Gifford AL, Rabeneck L, Zackin R, Sinclair G, Weissman S, Neidig J, Marcus C, Chesney M, Cohn SE, Wu AW; Adult AIDS Clinical Trials Unit Outcomes Committee. Development and validation of a self-completed HIV symptom index. J Clin Epidemiol. 2001 Dec;54 Suppl 1:S77-90. doi: 10.1016/s0895-4356(01)00449-8. PMID 11750213
- See also: SF-36® Health Survey Update by John E. Ware, Jr., Ph.D. — http://www.sf-36.org/tools/sf36.shtml